CLINICAL TRIAL: NCT04637971
Title: Coaching Intervention to Improve Mental Well-being of Community Women Who Are At-risk for Common Mental Disorders in Hong Kong: a Randomised Controlled Trial
Brief Title: Coaching Intervention in Women At-risk for Common Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yi-Nam Suen, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iCMD_Coaching_RCT
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Common Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching (Experimental): The present intervention is a structured, group-based coaching program that is facilitating an active process of change through the identification of achievable personal goals, the formulation of action plans, the provision of constructive feedback, and progressive monitoring of goal attainment.
  Interventions: Other: Coaching
- Self-help tips plus telephone support (Active Comparator): Self-help tips including stress coping methods. Our project staff will contact the subject to encourage her to make use of the tips we sent her.
  Interventions: Other: Self-help tips plus telephone support

INTERVENTIONS:
Other: Coaching — Participants will receive 4 sessions of group coaching intervention within 6 weeks. Each session is in a group of 3-4 women and lasts for approximately 1.5 hours. The sessions will be conducted by experienced social workers.
  Arms: Coaching
Other: Self-help tips plus telephone support — Participants will receive 4 self-help tips sent via SMS and 4 phone call from a social worker in 6-week of time. During the telephone call, the social worker will advise the client to make use of the tips we sent to her.
  Arms: Self-help tips plus telephone support

SUMMARY:
This study aims to provide coaching intervention for prevention of developing common mental disorders to 60 at-risk women in Hong Kong.

DETAILED DESCRIPTION:
Participants will be recruited through online screening tool. Eligible subjects with informed consent provided will be randomly assigned to coaching group or self-help tips plus telephone support group.

To test the effectiveness of the coaching intervention, data collection will be conducted on demographics, symptoms and psychosocial aspects at baseline, immediately, 3-month and 12-month post-intervention. A self-reported brief questionnaire will be administered at every intervention as well.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Able to understand Cantonese and read/write Chinese
* With subsyndromal or minor common mental disorders (CMD) indicated by 10 - 20 of Depression subscale of Depression, Anxiety and Stress Scale (DASS) or 8-14 of Anxiety subscale of DASS

Exclusion Criteria:

* Those mental conditions that require other treatment priorities (e.g., suicidal risk, substance abuse, current or past episodes of psychotic disorder, personality disorders)
* Those medical conditions that severely limit participation, comprehension, or adherence to treatment (e.g., epilepsy, dementia, terminal medical illness)
* Those who are receiving structured psychotherapy or counseling

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms | 6-month post-intervention
  Score of depression subscale of Depression, Anxiety and Stress Scale (DASS) at 6-month post-intervention will be compared with that at baseline.
Changes in anxiety symptoms | 6-month post-intervention
  Score of anxiety subscale of Depression, Anxiety and Stress Scale (DASS) at 6-month post-intervention will be compared with that at baseline.

SECONDARY OUTCOMES:
Changes in depressive symptoms | Immediate and 3-month post-intervention
  Score of depression subscale of Depression, Anxiety and Stress Scale (DASS) immediate and 3-month post-intervention will be compared with that at baseline.
Changes in anxiety symptoms | Immediate and 3-month post-intervention
  Score of anxiety subscale of Depression, Anxiety and Stress Scale (DASS) immediate and 3-month post-intervention will be compared with that at baseline.
Changes in quality of life | Immediate, 3- and 6-month post-intervention
  Score of 12-Item Short Form Health Survey version 2 (SF-12 v2) immediate, 3- and 6-month post-intervention will be compared with that at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Nam Suen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No